CLINICAL TRIAL: NCT06134063
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study on the Efficacy and Safety of Xuanfei Baidu Granule in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Study on the Efficacy and Safety of Xuanfei Baidu Granule in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Cuiling Feng, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XFBD-AECOPD-001
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Xuanfei Baidu granule

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Xuanfei Baidu granule
- Control group (Placebo Comparator)
  Interventions: Drug: Xuanfei Baidu granule Placebo

INTERVENTIONS:
Drug: Xuanfei Baidu granule — Xuanfei Baidu granule will be administered twice daily for 7 days on the basis of basic treatment
  Arms: Experimental group
Drug: Xuanfei Baidu granule Placebo — Xuanfei Baidu granule Placebo will be administered twice daily for 7 days on the basis of basic treatment
  Arms: Control group

SUMMARY:
This study is a prospective,multicenter, randomized, double-blind, placebo-controlled trial.

This study plans to enroll 375 participants who will be randomly assigned in a 2:1 ratio. On the basis of basic treatment, one group will receive Xuanfei Baidu granule, while the other group will receive Xuanfei Baidu granule placebo, with one sachet in the morning and one in the evening, for a duration of 7 days. Visits will be conducted on days 7, 14, and 21 after enrollment.

If any participant experiences an acute exacerbation of chronic obstructive pulmonary disease (COPD) requiring hospitalization during the treatment period, they will continue taking the medication until the 7-day course is completed. In case of a COPD exacerbation hospitalization event during the study, hospital admission date, duration of hospitalization, and the treatment regimen during hospitalization will be recorded.

DETAILED DESCRIPTION:
This study is a prospective,multicenter, randomized, double-blind, placebo-controlled trial.

This study plans to enroll 375 participants who will be randomly assigned in a 2:1 ratio. On the basis of basic treatment, one group will receive Xuanfei Baidu granule, while the other group will receive Xuanfei Baidu granule placebo, with one sachet in the morning and one in the evening, for a duration of 7 days. Visits will be conducted on days 7, 14, and 21 after enrollment.

If any participant experiences an acute exacerbation of chronic obstructive pulmonary disease (COPD) requiring hospitalization during the treatment period, they will continue taking the medication until the 7-day course is completed. In case of a COPD exacerbation hospitalization event during the study, hospital admission date, duration of hospitalization, and the treatment regimen during hospitalization will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 80 years old, including 40 and 80 years old, regardless of gender;
* Clinical records of traceable of the chronic obstructive pulmonary disease history records, after bronchodilator FEV1 less than 80% of the expected value;
* Comply with the definition of COPD acute exacerbations and with mild and moderate severity assessment;
* Symptoms of AECOPD time less than 48 h;
* "Shiduyufei" diagnostic standard;
* Volunteered for the study, signed informed consent, is willing to cooperate with the visitor.

Exclusion Criteria:

* Patients showing signs of hospitalization;
* With respiratory system diseases other than the AECOPD (for example, pneumonia, bronchiectasis, active tuberculosis, pneumothorax, pleural effusion, pulmonary embolism, or affect the respiratory movement function of neuromuscular diseases, etc.);
* Patients with severe basic diseases (for example, uncontrolled hypertension diabetes and complicated with heart failure (NYHA class IV), severe arrhythmia, acute coronary syndrome, hemodynamic instability, long-term use of immunosuppressive agents, etc.);
* With primary disease such as tumor or blood system;
* With severe liver disease (cirrhosis, portal hypertension, varices bleeding) or renal insufficiency;
* Pregnant women and breastfeeding mothers, those suspected of being pregnant, or women of childbearing age at risk of pregnancy who have not taken effective contraceptive measures;
* Dementia, mental disorders, such as unable to read or understand the research content, the information collection;
* With drug allergy;
* 3 months prior to screening for other interventional clinical research and the research data information;
* Within 1 week before screening been oral Chinese medicine or other proprietary Chinese medicine treatment;
* Patient refused to sign a consent form, or estimate adherence is poor, or follow-up possibilities is poor.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate. | within 21 days after enrollment
  Admission for acute exacerbation of COPD within 21 days after enrollment (excluding admission for reimbursement).

SECONDARY OUTCOMES:
Duration of acute exacerbation of COPD in this episode. | within 21 days after enrollment
  Duration of acute exacerbation of COPD in this episode.
Change in the Dyspnea Visual Analog Scale (VAS) score after treatment compared to baseline: Assessing the severity of breathlessness on days 7, 14, and 21 after enrollment. | days 7, 14, and 21 after enrollment
  The minimum and maximum values for VAS scores are 0 and 10. A higher score indicates a worse outcome.
Change in the COPD Assessment Test (CAT) score after treatment compared to baseline: Assessing the degree of health impairment on days 7, 14, and 21 after enrollment. | on days 7, 14, and 21 after enrollment
  The CAT score ranges from 0 to 40. Patients scoring 0 to 10 points are classified as having "mild impact" of COPD, 11 to 20 points as "moderate impact," 21 to 30 points as "severe impact," and 31 to 40 points as "very severe impact.
Change in the mMRC score after treatment compared to baseline: Assessing the severity of breathlessness on days 7, 14, and 21 after enrollment. | on days 7, 14, and 21 after enrollment
  The minimum and maximum values for mMRC scores are 0 and 4. A higher score indicates a worse outcome.
  Grade 0 means I only get breathless with strenuous exercise; Grade 1 means I get short of breath when hurrying on the level or walking up a slight hill; Grade 2 means I walk slower than people of the same age on the level because of breathlessness, or I have to stop for rest when walking at my own pace on the level; Grade 3 means I stop for breath after walking about 100 meters or after a few minutes on the level; Grade 4 means I am too breathless to leave the house or I am breathless when dressing or undressing.
Change in the Exacerbations of Chronic Pulmonary Disease Tool (EXACT) score after treatment compared to baseline: Assessing daily COPD exacerbation events within 21 days after enrollment. | within 21 days after enrollment
  The minimum and maximum values for EXACT scores are 0 and 70. A higher score indicates a worse outcome.
Change in the Clinical Symptom Score after treatment compared to baseline: Observing clinical symptom scores on days 7, 14, and 21 after enrollment. | on days 7, 14, and 21 after enrollment
  The clinical symptom score is based on the individual symptoms of the patient graded as none, mild, moderate, or severe, with scores of 0, 1, 2, and 3, respectively. The scores for each individual symptom are then added up to obtain the total score, ranging from a minimum of 0 to a maximum of 27. A higher total score indicates a more severe outcome.
Incidence of clinical abnormalities in laboratory examination and electrocardiogram. | within 21 days after enrollment
  Incidence of clinical abnormalities in laboratory examination and electrocardiogram.
Incidence of adverse events and serious adverse events. | within 21 days after enrollment
  Incidence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China